CLINICAL TRIAL: NCT01355614
Title: A Multi-center, Randomized, Double-blind, Active Controlled Study to Assess Efficacy, Safety and Tolerability of the Anti-IL13 Monoclonal Antibody QAX576 in the Treatment of Perianal Fistulas in Patients Suffering From Crohn's Disease
Brief Title: A Phase II Efficacy Study in Fistulizing Crohn's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAX576A2209; 2010-019973-13 (EudraCT Number)
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Fistula
MeSH Terms: conditions — Crohn Disease; Fistula | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- QAX576 (Experimental)
  Interventions: Drug: QAX576
- Infliximab (Other)
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: QAX576
  Arms: QAX576
Drug: Infliximab
  Arms: Infliximab

SUMMARY:
This study will assess the safety and efficacy of QAX576 if patients with fistulizing Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* At least one draining enterocutaneous perianal fistula
* Diagnosis of Crohn's disease (CD) must have been established for at least 6 months
* At least one ineffective fistula treatment (but no previously failed anti-TNFα (tumour necrosis factor) antibody treatment)
* Patients should not suffer from any other health problems that may jeopardize their participation in the study.

Exclusion Criteria:

* Current or recent (within 30 days of enrollment, or 5 half-lives of the compound, whichever is longer) use of anti-TNFα antibody treatment
* Active Crohn's disease
* Recent or pending abdominal or ano-rectal surgery, particularly presence of stricture, or abscess, or retention for which surgery might be indicated
* Previously failed anti-TNFα antibody treatment
* Intercurrent bacterial or viral (intestinal) infection (serologically or microbiologically confirmed)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy of QAX576 to induce complete closure for at least 4 weeks of all perianal fistulas in patients suffering from Crohn's disease by: clinical observation and cutaneous photodocumentation | 52 weeks

SECONDARY OUTCOMES:
Assessment of safety and tolerability of QAX576 in patients suffering from Crohn's disease as measured by lab assessments, ECG, physical exam etc | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Germany (5):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Kiel, Germany
  - Novartis Investigative Site, München, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Jena
- Novartis Investigative Site, Zurich, Switzerland

REFERENCES:
- See also: Results for CQAX576A2209 from the Novartis Results Repository — http://oak.novartis.com/21363/